CLINICAL TRIAL: NCT04143529
Title: Preoperative Mindfulness in Musculoskeletal Tumor Patients
Brief Title: Preoperative Mindfulness In Musculoskeletal Tumor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Prinicipal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-097
Record Dates: First submitted 2019-08-27; First posted 2019-10-29 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Musculoskeletal Malignancy
Keywords: Musculoskeletal malignancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized acceptance-based mindfulness exercise (Experimental): The purpose of this study is to identify whether a brief 60-second acceptance based mindfulness intervention at specific time points will reduce state trait anxiety, Mini-Mental Adjustment to Cancer Scale score, pain intensity, distress, anxiety, depression and anger
  Interventions: Behavioral: Personalized acceptance-based mindfulness exercise
- Brief educational pamphlet (Placebo Comparator): The control condition will be educational information on pain and stress that patients will read over within 60 second at specific timepoints.
  Interventions: Behavioral: Brief educational pamphlet

INTERVENTIONS:
Behavioral: Personalized acceptance-based mindfulness exercise — The mindfulness intervention will be a video-flash found at http://www.pixelthoughts.co. In this exercise patients are asked to write down a concern or worry, and watch it get put into perspective within a 60 seconds time frame.
  Arms: Personalized acceptance-based mindfulness exercise
Behavioral: Brief educational pamphlet — The control condition will be educational information on pain and stress that patients will read over within 60 seconds
  Arms: Brief educational pamphlet

SUMMARY:
Psychosocial distress is common in patients with an oncologic diagnosis, with anxiety being present in almost 20-30% of the patients.[1, 2, 10] Mindfulness exercises have shown to reduce this distress.[4, 5]

Recently, the implementation of a 60-second mindfulness-based intervention has shown to have momentary effects on pain, anxiety, depression and anger in orthopaedic upper extremity patients.[9] However, its lasting effect after the single intervention was not evaluated. Nonetheless, because the intervention is not time consuming and is easy to implement it may benefit orthopaedic oncology patients in their pre-operative coping.

The implementation of a 60-second mindfulness-based intervention has shown to have momentary effects on pain, anxiety, depression and anger in orthopaedic upper extremity participants. In this research study, the investigators are studying a 60-second interactive personalized acceptance-based mindfulness exercise

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of a preoperative 60-second interactive personalized acceptance-based mindfulness exercise (intervention) versus a brief educational pamphlet (control) on anxiety in patients undergoing curative surgery for a musculoskeletal malignancy.

ELIGIBILITY:
Inclusion Criteria:

* All adult (>18 years) patients attending the Orthopaedic Oncology Department outpatient clinic (Dr. Santiago Lozano-Calderon, Dr. Kevin Raskin, Dr. J. Schwab) at the MGH with a histologically confirmed musculoskeletal malignancy undergoing curative surgery will be enrolled at their last preoperative visit.

  * Patients with a musculoskeletal malignancy undergoing curative surgical treatment
  * Histologic confirmation of malignancy prior to curative surgery
  * Primary surgery of musculoskeletal malignancy at the Massachusetts General Hospital
  * Able to give informed consent
  * English fluency and literacy

    --- English fluency is needed because the intervention (a 60-seconds video) is in English and there is no alternate version available.
  * Age ≥18 years

Exclusion criteria:

* Significant axis I or II psychopathology that would interfere with participation in the study
* Pregnant patients
* Metastasis at presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Difference in State Trait Anxiety Score between Groups | from enrollment to the day of admission for surgery up to 3 weeks
  State-Trait Anxiety Inventory (STAI) for Adults - Form Y-1, is a measure to evaluate trait and state anxiety and helps to diagnose anxiety and to differentiate it from depressive syndromes

SECONDARY OUTCOMES:
Difference in Pain Intensity Score between Groups | from enrollment to the day of admission for surgery up to 3 weeks
  Pain Intensity as measured by Ordinal rating of Pain (0-10), this will allow us to measure changes in pain amongst subjects
Difference in Distress Score between Groups | from enrollment to the day of admission for surgery up to 3 weeks
  Mini-Mental Adjustment to Cancer Scale which evaluates the coping across four strategies: anxious preoccupation, fighting spirit, helplessness-hopelessness and positive redefinition.
Difference in Anxiety Score between Groups | from enrollment to the day of admission for surgery up to 3 weeks
  Mini-Mental Adjustment to Cancer Scale which evaluates the coping across four strategies: anxious preoccupation, fighting spirit, helplessness-hopelessness and positive redefinition.
Difference in Depression Score between Groups | from enrollment to the day of admission for surgery up to 3 weeks
  Mini-Mental Adjustment to Cancer Scale which evaluates the coping across four strategies: anxious preoccupation, fighting spirit, helplessness-hopelessness and positive redefinition.
Difference in Anger Score between Groups | from enrollment to the day of admission for surgery up to 3 weeks
  Mini-Mental Adjustment to Cancer Scale which evaluates the coping across four strategies: anxious preoccupation, fighting spirit, helplessness-hopelessness and positive redefinition.

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation
URL: http://www.partners.org/innovation